CLINICAL TRIAL: NCT00536406
Title: BE-ACTIV: Treating Depression in Nursing Homes
Brief Title: Evaluating a Behavioral Activities Treatment Program for Depressed Nursing Home Residents
Acronym: BE-ACTIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Suzanne Meeks, Principal Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH074865 (NIH); R01MH074865 (NIH); DATR A4-GPS
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: Geriatric; Nursing Homes
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Participants will receive the BE-ACTIV treatment
  Interventions: Behavioral: BE-ACTIV
- B (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: BE-ACTIV — BE-ACTIV is 10-week behavioral treatment involving increasing pleasant events.
  Arms: A
Behavioral: Treatment as usual (TAU) — TAU includes usual treatment in nursing care facility.
  Arms: B

SUMMARY:
This study will evaluate whether a behavioral activities treatment program improves symptoms of depression in nursing home residents.

DETAILED DESCRIPTION:
Depression is a common mental disorder that affects nearly half of all older people living in nursing homes. Depression can severely impact people's lives, causing them to often feel sad and hopeless, as well as affect people's sleep patterns, concentration, and energy levels. In addition, nursing homes are often understaffed and very busy, making it difficult for older people with depression to receive a proper diagnosis and adequate treatment. Recent studies have shown that an increase in pleasurable activities among residents in nursing homes can improve symptoms of depression. The purpose of this study is to determine whether symptoms of depression can be reduced by increasing opportunities for nursing home residents to engage in pleasant events and build better relationships with nursing home staff members.

Participating nursing homes will be randomly assigned to have their residents receive behavioral activity treatment (BE-ACTIV) or treatment as usual for 12 weeks. Potential participating nursing home residents will complete two brief tests regarding memory, attention, and symptoms of depression. An hour-long interview will then be conducted during which eligible participating residents will discuss their symptoms of depression, rate their health and level of functioning, and assess the quality of their relationship with a staff member. Residents receiving BE-ACTIV will meet with a therapist for weekly 30-minute sessions for 10 weeks. During these sessions, residents will discuss their activity participation and any pleasant events that they recently experienced. Therapists and nursing home activities staff will work together to incorporate more activities of interest into each resident's schedule. Residents of nursing homes assigned to receive treatment as usual will be asked to rate their mood once a week for 10 weeks. Researchers will observe each resident, regardless of treatment group, for 5-minute intervals at various times during the study to assess mood and activity levels. All participating residents will undergo a second interview after 10 weeks to discuss any changes or improvements in mood, symptoms of depression, activity level, or their relationship with staff members. All participating residents will be assessed after 3 months and again after 6 months post-treatment to determine whether the BE-ACTIV program was successful in improving symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents in long-term care beds with an expected stay of 3 months or more
* Geriatric Depression Scale score of at least 11
* Meets DSM-IV criteria for major depressive disorder or research diagnostic criteria for minor depressive disorder

Exclusion Criteria:

* Mini Mental State Exam score below 14
* Referred to hospice care for a terminal condition
* Current unstable or terminal medical condition
* Suicidal
* Meets DSM-IV criteria for bipolar disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-08; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Depression diagnosis and depressive symptoms as assessed by the Geriatric Depression Scale | Measured at Weeks 12, 24, and 48
Functioning as assessed by the Dartmouth COOP Scales for Social Functioning | Measured at Weeks 12, 24, and 48

SECONDARY OUTCOMES:
Staff attention | Measured at Weeks 12, 24, and 48
Positive affect | Measured at Weeks 12, 24, and 48
Activity participation | Measured at Weeks 12, 24, and 48
Behavior problems | Measured at Weeks 12, 24, and 48
Resident satisfaction | Measured at Weeks 12, 24, and 48

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Meeks, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States